CLINICAL TRIAL: NCT04885907
Title: A Randomised, Blinded, Controlled Trial of a Third Dose of Moderna COVID-19 Vaccine Versus Placebo in Solid Organ Transplant Recipients
Brief Title: Third Dose of Moderna COVID-19 Vaccine in Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Deepali Kumar, Clinician-Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-5324.0
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Vaccine Response Impaired; Immune Suppression; Covid19
Keywords: solid organ transplant; vaccine
MeSH Terms: conditions — COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Intervention Model Description: Randomised, placebo-controlled trial
Who Masked: Participant, Care Provider
Masking Description: Participant and vaccinator will be blinded to vaccine vs placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental group (Active Comparator): Participants will receive a one dose of mRNA-1273 vaccine 0.5mL i.m. in deltoid muscle
  Interventions: Biological: mRNA-1273 vaccine
- Comparator Group (Placebo Comparator): Participants will receive one dose of normal saline injection 0.5mL i.m. in deltoid muscle
  Interventions: Other: Normal Saline Placebo

INTERVENTIONS:
Biological: mRNA-1273 vaccine — COVID vaccine 3rd dose
  Other Names: Moderna COVID-19 vaccine
  Arms: Experimental group
Other: Normal Saline Placebo — Normal Saline Placebo
  Arms: Comparator Group

SUMMARY:
This study will be a randomized, double-blind, placebo-controlled trial of a third dose of Moderna vaccine versus placebo. Participants will be those that have received two doses of mRNA-1273 COVID vaccine (Moderna) at 0 and 1 months. Participants will be randomized 1:1 to receive either a third dose of the mRNA-1273 vaccine or saline placebo at 3 months post initial vaccination.

DETAILED DESCRIPTION:
Solid organ transplant (SOT) recipients are at high risk of COVID-19 complications. The Moderna vaccine (mRNA-1273) has proven highly efficacious and safe in a phase III large, randomized controlled trial of 30,420 persons in the general population, and has been in use in Canada since December 2020. SOT patients show diminished response to mRNA vaccines in several studies with approximately 40-50% positive antibody after the second dose. In positive patients, antibody titers are lower than the general population and adverse events mirror the general population. The current study will recruit 120 SOT recipients who have received both scheduled doses of the Moderna vaccine at 0 and 1 months. The hypothesis is that a third dose of vaccine will significantly increase antibody titers. SOT participants will be recruited and randomized 1:1 to receive an additional dose of Moderna COVID-19 vaccine two months after the last dose vs saline placebo. The outcomes will measure anti-RBD antibody titer, T-cell immunity, local/systemic side effects, and rejection events.

ELIGIBILITY:
Inclusion Criteria:

* Solid organ transplant recipient who has previously received Moderna vaccine at 0 and 1 months
* Able to provide informed consent

Exclusion Criteria:

* Anaphylaxis or allergic reaction to Moderna vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
anti-RBD antibody titer | 4-6 weeks after intervention
  Percentage of patients that achieve anti-RBD of >=100 U/mL in each arm

SECONDARY OUTCOMES:
Adverse events | 7 days after intervention
  Percentage of patient with local and systemic adverse events
T-cell response | 4-6 weeks after intervention
  Proportion of participants with an increase in polyfunctional T-cell response compared to pre-vaccination

OTHER OUTCOMES:
SARS-CoV-2 infection | 6 months after intervention
  Number of patients with microbiologically proven infection
Rejection | 4 weeks after intervention
  Proportion of patients with biopsy-proven or clinically treated graft rejection

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, MD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - University Health Network, Toronto General Hospital, Toronto, Ontario
  - University Health Network, Toronto General Hospital, Multi-Organ Transplant, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baden LR, El Sahly HM, Essink B, Kotloff K, Frey S, Novak R, Diemert D, Spector SA, Rouphael N, Creech CB, McGettigan J, Khetan S, Segall N, Solis J, Brosz A, Fierro C, Schwartz H, Neuzil K, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Mascola J, Polakowski L, Ledgerwood J, Graham BS, Bennett H, Pajon R, Knightly C, Leav B, Deng W, Zhou H, Han S, Ivarsson M, Miller J, Zaks T; COVE Study Group. Efficacy and Safety of the mRNA-1273 SARS-CoV-2 Vaccine. N Engl J Med. 2021 Feb 4;384(5):403-416. doi: 10.1056/NEJMoa2035389. Epub 2020 Dec 30. PMID 33378609
- [Derived] Kumar D, Ferreira VH, Hall VG, Hu Q, Samson R, Ku T, Ierullo M, Majchrzak-Kita B, Tomlinson G, Gingras AC, Humar A. Neutralization of SARS-CoV-2 Variants in Transplant Recipients After Two and Three Doses of mRNA-1273 Vaccine : Secondary Analysis of a Randomized Trial. Ann Intern Med. 2022 Feb;175(2):226-233. doi: 10.7326/M21-3480. Epub 2021 Nov 23. PMID 34807716